CLINICAL TRIAL: NCT07075029
Title: RSV in Acute Respiratory Infection Surveillance Among Community-Dwelling Elderly Aged ≥50 Years in China: A Prospective, Observational, Community-Based Study
Brief Title: RSV in Acute Respiratory Infection Surveillance Among Community-Dwelling Elderly Aged ≥50 Years in China
Acronym: RAISE
Status: Not yet recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Huashen Institute of Microbes and Infections (Unknown)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases Affiliation, Huashan Hospital; Shanghai Huashen Institute of Microbes and Infections, Huashan Hospital
Other Study IDs: RAISE
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Acute Respiratory Infections (ARIs)
Keywords: RSV; Acute Respiratory Infections; Community

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRE-ARI group: CRE-ARI group will includes individuals aged 50 years and older who self-report symptoms of acute respiratory infection (ARI) to the investigators/study personnel during the study period.
  Interventions: Diagnostic Test: NP swabs
- CAI group: Cohabitants of individuals with ARI will also be enrolled in the study, forming the Cohabitants of ARI Individuals (CAI) group. Eligible participants in this group include older adults aged ≥50 years and children under 5 years of age.
  Interventions: Diagnostic Test: NP swabs

INTERVENTIONS:
Diagnostic Test: NP swabs — Nasopharyngeal (NP) swabs will be collected from all participants for respiratory pathogen detection using point-of-care testing (POCT) and/or centralized laboratory analysis.

SUMMARY:
This is a multicenter, prospective, observational, community-based study designed to evaluate the incidence of respiratory syncytial virus (RSV) infection among community-dwelling elderly individuals in China, as well as their cohabiting older adults and children, over a 24-month period. During the study, home visits will be conducted to collect nasopharyngeal (NP) swabs from all community residents aged ≥50 years who report symptoms of acute respiratory infection (ARI). Pathogen detection will be performed using both point-of-care testing (POCT) and centralized laboratory analysis.

DETAILED DESCRIPTION:
The study will cover about 10 communities representing diverse geographical locations, economic conditions, and population densities.

ELIGIBILITY:
Inclusion Criteria:

* CRE-ARI group:

  1. Male or female adults aged ≥50 years (calculated based on date of birth and date of visit).
  2. Presence one of the following conditions of ARI case definition :

     * At least two respiratory symptoms/signs within 48 hours prior to self-reporting OR
     * At least one respiratory symptom/sign + one systemic symptom/sign within 48 hours prior to self-reporting
  3. Provision of written informed consent by the participant or their legal guardian, in accordance with local EC (Ethics Committee) requirements.
* CAI group:

  1. In the household, include at least one patient meeting the inclusion criteria (index case[s]) of CRE-ARI group.
  2. Male or female adults aged ≥50 years or children aged<5 years (calculated based on date of birth and date of visit).
  3. In the household, apart from the index case(s), there are two or more members who meet the criteria (2) AND are willing to participate, regardless of whether these household members exhibit ARI symptoms.
  4. Provision of written informed consent by the participant or their legal guardian, in accordance with local EC (Ethics Committee) requirements.

Exclusion Criteria:

1. Enrollment in the CRE-ARI group within the preceding 14 days.
2. Enrollment in the CRE-ARI group has been more than 4 times during the previous 12 months (applicable only to the CRE-ARI group enrollment).
3. For CAI group, if a household has been enrolled into CAI group within the previous 12 months.
4. Residence outside the designated study catchment area.
5. Unwilling to provide consent/assent (if applicable) to participate.
6. Unwilling to provide biological samples.
7. Any other situation deemed inappropriate for participation by the investigator, including potential risks to the subject upon enrollment or factors that may affect the interpretation of study results, such as clinical judgment, safety concerns, or the integrity of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will cover approximately 10 communities. All individuals aged 50 years and older residing in these communities will be considered potential participants. Those who self-report symptoms of acute respiratory infection (ARI) will be enrolled. In addition, if their cohabitants meet the inclusion criteria, they will be enrolled as a family unit.
Sampling Method: Non-Probability Sample
Enrollment: 28800 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of RSV | From September 2025 to September 2027
  To investigate the incidence rate of RSV related acute respiratory infection (ARI) in community-dwelling adults of 50 years or older in China.

SECONDARY OUTCOMES:
Positive rate of RSV | From September 2025 to September 2027.
  To investigate the positive rate of RSV in the community-dwelling adults of 50 years or older with ARI in China.
Prevalence | From September 2025 to September 2027.
  To investigate the prevalence of common upper respiratory system infection pathogens in community-dwelling adults aged 50 years or older with ARI in China.
Association between symptoms and pathogens | From enrollment to the final sample collection on Day 7.
  To investigate the association between symptoms and pathogens in community-dwelling adults aged 50 years or older with ARIs through questionnaires. Symptoms include respiratory signs and symptoms, such as those related to upper and lower respiratory tract disease (URTD and LRTD), as well as systemic signs and symptoms.

OTHER OUTCOMES:
Assessment of risk and protective factors for RSV infection through questionnaires | From September 2025 to September 2027.
  To explore risk and protective factors for RSV infection in community-dwelling adults aged 50 years or older with ARI. Information on potential risk and protective factors, such as smoking status, household size, and out-of-home activity patterns, will be collected through questionnaires.
Association between symptoms and pathogens in high risk household members | From enrollment to the final sample collection on Day 7.
  To explore the association between symptoms and pathogens in high risk household members (age ≥50 years or <5 years) living together with community-dwelling ARI adults of 50 years or older through questionnaires. Symptoms include respiratory signs and symptoms, such as those related to upper and lower respiratory tract disease (URTD and LRTD), as well as systemic signs and symptoms.
Prevalence | From September 2025 to September 2027.
  To explore the prevalence of common upper respiratory system infection pathogen in high risk household members (age ≥50 years or <5 years) living with community-dwelling ARI adults of 50 years or older.
Healthcare seeking behaviors through questionnaires | From enrollment to the final sample collection on Day 7.
  To explore healthcare-seeking behaviors among community-dwelling adults aged 50 years or older with ARI through questionnaires. Healthcare-seeking behaviors include whether medical care was sought, adherence to medical advice versus self-medication, and the types of medications used.
Transmission of RSV | From enrollment to the final sample collection on Day 7.
  To explore RSV transmission among high-risk household members (aged ≥50 years or <5 years) living with community-dwelling ARI adults aged 50 years or older, through analysis of full-length RSV genomes from RSV-positive specimens. Sequencing data will be mapped, and candidate single nucleotide polymorphisms (SNPs) will be identified for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, MD, Principal Investigator — Huashan Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - The Third People's Hospital of Yichang, Yichang, Hubei
  - Nanjing Municipal Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - First People's Hospital of Jiujiang, Jiujiang, Jiangxi
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Affiliated Hospital of Yan'an University, Yanan, Shanxi
  - Baihe Town Community Health Service Center, Shanghai
  - Chinese People's Armed Police Force Characteristic Medical Center, Tianjing

IPD SHARING:
Plan to Share IPD: Undecided
After thesis defense the study may be published internationally to be available for the public.